CLINICAL TRIAL: NCT04976920
Title: Non-selection Trial Comparing Metabolomics to PGT-A Embryo Selection Using Vitrolife G-TL Media
Brief Title: Metabolomics Non Selection Study - Vitrolife Media
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Overture Life (Industry)
Collaborators: Clinica Juana Crespo (Unknown); Grupo Procrearte (Unknown)
Responsible Party: Principal Investigator, Dr. Jose Horcajadas, Principal Investigator, Overture Life
Other Study IDs: OLM001
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Infertility
Keywords: IVF; genetic screening; preimplantation genetic testing
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Patients will undergo a routine IVF cycle. This will include ovarian stimulation, egg retrieval and fertilization of oocytes through intracytoplasmic sperm injection (ICSI). All fertilized oocytes will be cultured up to blastocyst for five to six days.
  Spent media will be collected on day 5-6 for all embryos reaching blastocyst on day 5, and on day 6 for those reaching blastocyst on day 6. The spent culture media will be sent to a lab for metabolomic analysis.
  For the embryo transfer, the best morphology blastocyst will be selected for transfer by the New Hope embryologist. The embryo transfer outcome will be compared to the metabolomics result to determine the NPV and PPV of metabolomics vs implantation.
  Interventions: Diagnostic Test: Overture Metabolomics Embryo Selection

INTERVENTIONS:
Diagnostic Test: Overture Metabolomics Embryo Selection — Patients will have their embryos selected for transfer based on morphology alone. The embryo transfer outcome will be compared to the metabolomics result to determine the NPV and PPV of metabolomics vs implantation.

SUMMARY:
In this study, study investigators will collect embryo culture media on day 5 of vitro fertilization (IVF) culture, prior to vitrification and embryo transfer for testing via Metabolomic screening. Metabolomics is a new, non-invasive method of embryo selection which involves testing discarded embryo culture media for analytes secreted by the developing embryo. These analytes can be used to determine the implantation potential, and ploidy, of the embryo.

DETAILED DESCRIPTION:
Patients will undergo a routine IVF cycle. This will include ovarian stimulation, egg retrieval and fertilization of oocytes through intracytoplasmic sperm injection (ICSI). All fertilized oocytes will be cultured up to blastocyst for five to six days.

Spent media will be collected on day 5-6 for all embryos reaching blastocyst on day 5, and on day 6 for those reaching blastocyst on day 6. The spent culture media will be sent to a lab for metabolomic analysis.

For the embryo transfer, the best morphology blastocyst will be selected for transfer by the New Hope embryologist.

Approximately 8-11 days after the embryo transfer, the patient will return to the clinic for a serum pregnancy test. Should the test be negative, they will be closed out of the study. Should the test be positive, they will continue to be monitored.

The patient will return to the clinic at approximately 8 weeks after embryo transfer for a serum pregnancy test, and an ultrasound to detect fetal heartbeat. The outcome will be documented and the patient closed out of the study at this time.

The embryo transfer outcome will be compared to the metabolomics result to determine the NPV and PPV of metabolomics vs implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age, 25% of patients <35 years, 25% of patients 35-37, 25% of patients 38-40, and 25% of patients >40 years.
* Signed Subject Consent Form. No inferior limit on number of eggs

Exclusion Criteria:

At the time of initial visit:

* Require or request PGT of any kind
* Low ovarian reserve defined as follicle stimulating hormone (FSH) >10 IU/L on day 2-4 of a prior menstrual cycle and anti-mullerian hormone (AMH) <15 pmol/L (or <2 ng/ml) within prior 12 months of cycle start

At the time of embryo selection:

-Patients without at least one embryo to transfer.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients recruited from an IVF center
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value (NPV) and positive predictive value (PPV) for MEI vs. expected implantation based solely on morphology. | Approximately 4-5 months, inclusive of IVF cycle, embryo transfer and monitoring up to eight weeks
  PPV (MEI high potential implanting / Total implanting), NPV (MEI low potential implanting / Total not implanting)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Horcajadas, PhD, Principal Investigator — Overture Life; Santiago Munne, PhD, Principal Investigator — Overture Life
Locations (2):
- Grupo Procrearte, Buenos Aires, Argentina
- Clinical Juana Crespo, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be presented at industry conferences, and published in peer reviewed journals.